CLINICAL TRIAL: NCT07190118
Title: Effects of Emicizumab Treatment on the Musculoskeletal System in Children With Hemophilia A: A Prospective Study
Brief Title: Effects of Emicizumab Treatment in Patients With Hemophilia A
Status: Not yet recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Asisst. Prof. Dr., Hasan Kalyoncu University
Other Study IDs: 2025/096
Record Dates: First submitted 2025-09-01; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A; Musculoskeletal Assessment; Musculoskeletal Abnormalities
Keywords: Hemophilia A; Emicizumab; Musculoskeletal system; Measurement
MeSH Terms: conditions — Hemophilia A; Musculoskeletal Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A Group: This will be the first assessment before the child begins treatment with emicizumab. During the first month of treatment, the child and parents will be asked to note any joint or muscle bleeding, including the bleeding site, duration of bleeding, and whether hospitalization is necessary. At the end of the first month, parents will be contacted by phone to assess bleeding episodes, and any bleeding that occurred during the first month will be recorded. The same assessments will then be repeated at the third and sixth months of treatment. The effectiveness of the treatment will be assessed after the first six months through an analysis of the assessments.

SUMMARY:
The aim of our study is to investigate the effects of emicizumab treatment on the musculoskeletal system in children with hemophilia A.

DETAILED DESCRIPTION:
Hemophilia is a rare inherited coagulation disorder resulting from a deficiency of factor (F) VIII or IX. It is a chronic group of diseases that primarily manifests as intra-articular (hemarthrosis) and intramuscular (hematoma) bleeding and affects quality of life. Easy ecchymosis formation in early childhood, especially spontaneous intra-articular and intramuscular bleeding, and a history of bleeding lasting longer than expected after interventions and trauma should raise the suspicion of hemophilia. The severity of bleeding findings is directly related to the degree of FVIII or FIX deficiency. While the clinical picture varies depending on the duration and frequency of bleeding, the severity of the disease is classified as severe (<1% IU dL-1), moderate (1%-5% IU dL-1), and mild (5%-40% IU dL-1). Hemophilia A occurs in 85% of the population (1 in 5,000 male births), while this rate is 15% in Hemophilia B (1 in 30,000 male births). Treatment of hemophilia is primarily divided into treatment of acute bleeding and prophylaxis. The primary goal in the treatment of acute bleeding is to achieve hemostasis within the first two hours after the onset of symptoms. Patients often recognize a bleeding episode by a tingling sensation or an "aura" before the bleeding begins. In such cases, factor replacement therapy should be administered immediately. In a patient presenting with severe acute bleeding, after determining the location and severity of the bleeding, factor VIII or factor IX and high-dose clotting factor concentrate (CFC) are administered. Factor concentrate doses should be 50 IU/kg factor VIII or 100-120 IU/kg factor IX. Even if bleeding slows or stops, CFC should be administered to maintain healing. Frequent measurement of factor levels should be performed to ensure that desired levels are maintained. Acetylsalicylic acid (ASA) and nonsteroidal anti-inflammatory drugs (NSAIDs) should be avoided during pain management due to their effects on platelet function and increased risk of bleeding. Prophylaxis treatment includes treating acute bleeding as well as replacing the missing factor in cases where there is no bleeding. Prophylactic treatment has many advantages. Prophylaxis is generally initiated at an early age to prevent and reduce the risk of joint bleeding and the development of hemophilic arthropathy. Dosing is personalized and adjusted according to the severity of bleeding. It protects joint health by reducing hemarthrosis episodes and reduces the need for joint surgical interventions. Prophylactic factor replacement in hemophilia treatment is administered two or three times a week via intravenous infusion. Emicizumab, one of the alternative pharmacological treatments developed in recent years, is a subcutaneous treatment method that provides patients with access to the medication within clinical and financial healthcare services in Turkey as of May 2025. Emicizumab, Fitusiran, and Concizumab, both inhibit natural anticoagulant pathways. With these subcutaneous treatments, injection frequency can vary depending on the molecule, but can be daily, weekly, or monthly. One of the most important advantages of these treatments is their effectiveness in the presence of alloantibodies, which are a significant cause of morbidity and mortality in hemophilia. Treatment features such as reduced injection frequency of factor replacements administered subcutaneously, eliminating the need for intravenous infusions, and increasing physical activity opportunities are thought to produce significant benefits affecting quality of life, in addition to controlling and preventing bleeding. Therefore, new drugs that promise less bleeding with fewer and more comfortable injections are quite attractive. It is believed that reduced bleeding will equally reduce musculoskeletal damage, support improved joint health, and increase the individual's level of functionality, resulting in improved quality of life by ensuring independence in daily life. Improved musculoskeletal health and independence in daily life will increase children's exercise habits. The positive contributions to the musculoskeletal system, such as increased overall muscle mass and maintenance of joint health, will also increase the effectiveness of physiotherapy programs. There are no other studies examining the effects of this newly introduced drug on the musculoskeletal system in children in Turkey. Therefore, the aim of our study was to investigate the effects of emicizumab treatment on the musculoskeletal system in children with hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Children who are under 18 years of age,
* Have been diagnosed with Hemophilia A by a physician,
* Have a factor level of 1% (IU) or less,
* Have inhibitors positive or negative,
* Have no obstacles to starting subcutaneous (emicizumab) treatment,
* Willing to participate in the study

Exclusion Criteria:

- Children with a history of cerebrovascular bleeding who present any neurological findings that would prevent participation in the study

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Because hemophilia A is an X-linked recessive disease, girls are carriers and boys are affected by the disease. Therefore, the study population consists of boys.
Study Population: Male patients under 18 years of age diagnosed with hemophilia A will constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
The pain | through of the study, average 6 months
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Hemophilia Joint Health Score (HJHS) | through of the study, average 6 months
  Hemophilia Joint H is a scoring system that targets the evaluation of three major joints (elbow, knee, and ankle). Consists of a total of 9 questions: 8 questions assessing joints and 1 question providing a global gait score. The hemophilia joint health score is calculated by assessing joint swelling, the longevity of the swelling, the presence of atrophy in the surrounding soft tissue, crepitus during active movement, loss of flexion or extension, pain, muscle strength, and the total global gait score. Hemophilia Joint Health Score values range from 0 to 124, with higher scores indicating poorer joint health.
Lower extremity functionality and mobility- 5-Time Sit-to-Go Test | through of the study, average 6 months
  The 5-time sit-to-stand test is scored based on the time (in seconds to the nearest decimal place) in which a patient can move from a sitting position to a standing position and back to a sitting position five times. At the beginning of the test, the test participant is instructed to sit in a chair with their back straight. They are also instructed to fold their arms across their chest. The test participant should then be instructed to sit and stand five times as quickly as possible. The shorter the time taken to complete the test, the better the test result.
Upper extremity functionality | through of the study, average 6 months
  The Questionnaire for Arm, Shoulder, and Hand Disabilities (Q-DASH) will be used to assess individuals' upper extremity functions. This questionnaire is a self-administered measurement tool with validated validity and reliability in Turkish. The questionnaire, consisting of 30 questions, assesses the individual's ability to perform functional activities (21 items), pain (5 items), and psychosocial aspects of the disease (4 items). The total score ranges from 0 to 100, with a higher score indicating better outcomes.
Static balance | through of the study, average 6 months
  The One-Legged Standing Test will be administered to assess patients' static balance. In the one-leg standing test, the subject will stand with their arms hanging at their sides and lift each lower extremity one leg at a time, measuring the duration of their stance. The time will be stopped if they reposition their supporting leg, touch the ground with their raised foot, or seek support from an observer or any other support.
Lower extremity functionality and mobility- 30-second Sit-to-Go Test | through of the study, average 6 months
  The 30-Second Chair Test is administered using a folding chair without arms. The chair, with rubber feet, is placed against a wall to prevent movement. The participant sits in the center of the chair, back straight, feet approximately shoulder-width apart and slightly behind the knees, with one foot slightly in front of the other to assist with balance. Arms are crossed at the wrists and held toward the chest. The participant is encouraged to perform as many complete poses as possible in 30 seconds. The participant is asked to sit fully between each pose. The tester, monitoring the participant's performance to ensure proper form, silently counts the number of each pose. The score is the total number of poses performed in the 30 seconds (more than half the poses by the end of 30 seconds are considered complete poses).
Lower extremity functionality and mobility- Timed Up-and-Go Test | through of the study, average 6 months
  The Timed Up and Go Test (TUG) is a quick and easy-to-administer clinical test that assesses an individual's basic mobility skills. The test involves the patient rising from a standard chair, walking a distance of 3 meters (10 feet), turning around, returning to the chair, and sitting down again. The time taken to complete this task is recorded in seconds.

SECONDARY OUTCOMES:
Fear of movement | through of the study, average 6 months
  The Tampa Kinesiophobia Scale will be used to assess patients' fear of movement. The questionnaire, which will be used to measure individuals' perspectives on movement and their fear aspects, consists of 17 questions with total scores ranging from 17 to 68. Tampa scores greater than 37 indicate a high degree of kinesiophobia.
Functional independence levels | through of the study, average 6 months
  The scoring system, categorized according to the International Classification of Functioning, Disability, and Health (ICF), was developed by considering activities that may be affected in the daily lives of hemophilia patients. Being a performance-based scale, it can be used in different languages. The scale consists of eight questions covering the subparameters of self-care, transfer, and locomotion. The self-care subparameter includes eating and hygiene, bathing and dressing; the transfer subparameter includes chair and squatting; and the locomotion subparameter includes walking, climbing and descending stairs (12-14 steps), and running. Activities are scored on a scale of 1 to 4, depending on the degree of independence. The minimum score is 8, and the maximum is 32. A high score indicates an individual's functional independence.
Children's Quality of Life | through of the study, average 6 months
  The Children's Quality of Life Inventory (PedsQL) will be used to assess patients' quality of life. The scale consists of both child and parent assessment forms and assesses four subscales: physical functioning, social functioning, school life, and emotional well-being. The scale, consisting of 5-point Likert-type questions, measures the child's quality of life based on their life experiences over the past week. Scores from each subscale range from 0 to 100. Higher scores indicate better quality of life, while lower scores indicate problems in the relevant area. The parent and child forms can be evaluated separately to obtain results from different perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba GÖNEN, Asisst. Prof. Dr., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poonnoose PM, Manigandan C, Thomas R, Shyamkumar NK, Kavitha ML, Bhattacharji S, Srivastava A. Functional Independence Score in Haemophilia: a new performance-based instrument to measure disability. Haemophilia. 2005 Nov;11(6):598-602. doi: 10.1111/j.1365-2516.2005.01142.x. PMID 16236109
- [Background] Kumban W, Amatachaya S, Emasithi A, Siritaratiwat W. Five-times-sit-to-stand test in children with cerebral palsy: reliability and concurrent validity. NeuroRehabilitation. 2013;32(1):9-15. doi: 10.3233/NRE-130818. PMID 23422454
- [Background] McLaughlin P, Morris R, Chowdary P. Investigating the relationship between the HJHS and HAL in routine clinical practice: A retrospective review. Haemophilia. 2018 Nov;24(6):988-994. doi: 10.1111/hae.13614. Epub 2018 Oct 8. PMID 30295404
- [Background] R CB, A TO, S PA, J CJ, F Q, J NM, Ja LP. Using the Hemophilia Joint Health Score for assessment of children: Reliability of the Spanish version. Physiother Theory Pract. 2019 Apr;35(4):341-347. doi: 10.1080/09593985.2018.1443356. Epub 2018 Feb 27. PMID 29485331
- [Background] Sun J, Hilliard PE, Feldman BM, Zourikian N, Chen L, Blanchette VS, Luke KH, Poon MC. Chinese Hemophilia Joint Health Score 2.1 reliability study. Haemophilia. 2014 May;20(3):435-40. doi: 10.1111/hae.12330. Epub 2013 Dec 16. PMID 24330460
- [Background] Hilliard P, Funk S, Zourikian N, Bergstrom BM, Bradley CS, McLimont M, Manco-Johnson M, Petrini P, van den Berg M, Feldman BM. Hemophilia joint health score reliability study. Haemophilia. 2006 Sep;12(5):518-25. doi: 10.1111/j.1365-2516.2006.01312.x. PMID 16919083
- [Background] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Background] Steen Carlsson K, Andersson E, Berntorp E. Preference-based valuation of treatment attributes in haemophilia A using web survey. Haemophilia. 2017 Nov;23(6):894-903. doi: 10.1111/hae.13322. Epub 2017 Aug 29. PMID 28851125
- [Background] Meeks SL, Batsuli G. Hemophilia and inhibitors: current treatment options and potential new therapeutic approaches. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):657-662. doi: 10.1182/asheducation-2016.1.657. PMID 27913543
- [Background] Franchini M, Mannucci PM. Non-factor replacement therapy for haemophilia: a current update. Blood Transfus. 2018 Sep;16(5):457-461. doi: 10.2450/2018.0272-17. Epub 2018 Feb 14. PMID 29517971
- [Background] Sahu S, Lata I, Singh S, Kumar M. Revisiting hemophilia management in acute medicine. J Emerg Trauma Shock. 2011 Apr;4(2):292-8. doi: 10.4103/0974-2700.82225. PMID 21769217
- [Background] Srivastava A, Brewer AK, Mauser-Bunschoten EP, Key NS, Kitchen S, Llinas A, Ludlam CA, Mahlangu JN, Mulder K, Poon MC, Street A; Treatment Guidelines Working Group on Behalf of The World Federation Of Hemophilia. Guidelines for the management of hemophilia. Haemophilia. 2013 Jan;19(1):e1-47. doi: 10.1111/j.1365-2516.2012.02909.x. Epub 2012 Jul 6. PMID 22776238
- [Background] Mehta P, Reddivari AKR. Hemophilia. 2023 Jun 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551607/ PMID 31869071
- [Background] Srivastava A, Santagostino E, Dougall A, Kitchen S, Sutherland M, Pipe SW, Carcao M, Mahlangu J, Ragni MV, Windyga J, Llinas A, Goddard NJ, Mohan R, Poonnoose PM, Feldman BM, Lewis SZ, van den Berg HM, Pierce GF; WFH Guidelines for the Management of Hemophilia panelists and co-authors. WFH Guidelines for the Management of Hemophilia, 3rd edition. Haemophilia. 2020 Aug;26 Suppl 6:1-158. doi: 10.1111/hae.14046. Epub 2020 Aug 3. No abstract available. PMID 32744769